CLINICAL TRIAL: NCT01848236
Title: Effects of Vitamin D Insufficiency in Man
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, John Adams, M.D., Professor, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adams VitD 01
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D2 (Experimental): Total of 500,000 IU vitamin D2 (50,000 IU twice weekly for 5 weeks)
  Interventions: Dietary Supplement: Vitamin D2
- Vitamin D3 (Experimental): Total of 500,000 IU vitamin D3 (50,000 IU twice weekly for 5 weeks)
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D2 — Ergocalciferol vitamin D2
  Arms: Vitamin D2
Dietary Supplement: Vitamin D3 — Cholecalciferol vitamin D2
  Arms: Vitamin D3

SUMMARY:
We would like to determine if vitamin D insufficiency exists in different ethnic groups, if it has an effect on bone mass and muscle function, if it has an impact on the function of the cells of the immune system, and if the functioning level of these systems can be improved by stabilizing the vitamin D levels to within normal limits.

DETAILED DESCRIPTION:
Vitamin D is a hormone that can either be made in the skin under the influence of sunlight or absorbed from the diet. Roughly 50% of the U.S. population suffers from an insufficiency of vitamin D and its more active metabolites. This defect can result in disorders in the bones, muscles and immune system. In humans, these disorders usually present themselves as decreased bone mass, decreased muscle strength and increased susceptibility to some infections, respectively.

Therefore, the purpose of this study is to:

1. determine, by use of skeletal and immune biomarkers in the blood and urine, whether vitamin D insufficiency exists in differently pigmented ethnic groups; skin pigmentation blocks vitamin D production in the skin;
2. determine whether the vitamin D status of the host has an impact on bone mass and muscle function;
3. ascertain whether the vitamin D status of the host has an impact on the function of cells of the immune system;
4. determine the effects of correction of vitamin insufficiency on the musculoskeletal and immune systems.

All tests are designed to gauge the state of the circulating and urine factors that contribute to overall calcium balance and/or imbalance. This will include screening for the presence or absence of active and latent infection with the agent that causes TB. If evidence of active TB is identified, one of the physician investigators in this study will inform the subject of the outcome of the screening test and this information will be reported to the California State Health Department.

Additionally, blood and related medical information will ultimately be stored in our UCLA Repository (Human Vitamin D Sample Bank) in the CTRC (Clinical Translational Research Center) in order to allow sharing of the cells with other approved researchers. The cells may be used for other future research related to the purposes described above.

We will enroll vitamin D-deficient subjects (African American, Hispanic and white) and vitamin D-sufficient matching controls against which to compare them. Deficient subjects will be randomized to receive a total of 500,000 IU of vitamin D2 or D3, at the standard replacement dose of vitamin 50,000 IU twice weekly for 5 weeks. Subjects will complete screening medical history, questionnaire, biochemical and DXA (if indicated for low bone mineral density) screening, and exam of muscle strength and/or back curvature (if indicated). Blood and urine will be collected to gauge the state of the circulating and urine factors that contribute to the subjects' overall calcium balance and/or imbalance, and to test for TB. After 5 weeks of vitamin D treatment, subjects will return for repeat testings. Subjects who are still vitamin D-deficient will undergo an additional 5-week regimen. Subjects for whom changes in bone mineral density and/or muscle strength are outcome measures will return one year later for repeat testing.

ELIGIBILITY:
Inclusion Criteria:

* 25D levels <30 ng/ml (Vitamin D sufficient) OR <20 ng/ml (Vitamin D deficient)
* At least 18 years of age

Exclusion Criteria:

* Hypercalcemia
* Hyperparathyroidism
* Hyperthyroidism
* Hypercalciuria
* Renal disease
* Intestinal malabsorption any disorder that places the subject at risk for developing hypercalcemia or hypercalciuria during standard vitamin D replacement therapy owing to the presence of underlying dysregulated vitamin D metabolism (e.g., sarcoidosis, TB, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change in serum 25D | 5 weeks

SECONDARY OUTCOMES:
Change in bone mineral density by biochemistry | 5 weeks
Change in muscle strength by exam | 5 weeks
Change in muscle strength by questionnaire | 5 weeks
Change in bone mineral density by DXA scan | 5 weeks
Change in fractional urinary calcium:creatinine excretion ratio | 5 weeks
Change in serum 1,25D | 5 weeks
Change in serum iPTH | 5 weeks
Change in serum bone biomarkers | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John S Adams, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Shieh A, Chun RF, Ma C, Witzel S, Meyer B, Rafison B, Swinkels L, Huijs T, Pepkowitz S, Holmquist B, Hewison M, Adams JS. Effects of High-Dose Vitamin D2 Versus D3 on Total and Free 25-Hydroxyvitamin D and Markers of Calcium Balance. J Clin Endocrinol Metab. 2016 Aug;101(8):3070-8. doi: 10.1210/jc.2016-1871. Epub 2016 May 18. PMID 27192696